CLINICAL TRIAL: NCT01509339
Title: Pharmacokinetics of Vancomycin for Inhalation in Cystic Fibrosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lab unable to measure vancomycin levels in Sputum
Sponsor: Case Western Reserve University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Elliott Dasenbrook, Assistant Professor of Medicine and Pediatrics, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iVCM 1.0
Record Dates: First submitted 2012-01-09; First posted 2012-01-13 (Estimated); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Cystic Fibrosis; Methicillin-resistant Staphylococcus Aureus
Keywords: Vancomycin; Inhalation; Nebulization; Pharmacokinetics
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Aspiration | interventions — Vancomycin; Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vancomycin for Inhalation (Experimental): 250 mg vancomycin in 5cc sterile water will be inhaled once. Patients will use a Pari Sprint nebulizer and Pari Vios compressor as the delivery system.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — 250 mg vancomycin in 5cc sterile water will be inhaled once. Patients will use a Pari Sprint nebulizer and Pari Vios compressor as the delivery system.
  Other Names: Nebulized vancomycin; Inhaled Vancomycin; Vancomycin for inhalation; Aerosolized Vancomycin

SUMMARY:
The purpose of this study is to determine the pharmacokinetics and safety of inhaled vancomycin in patients with cystic fibrosis.

DETAILED DESCRIPTION:
The prevalence of methicillin resistant Staphylococcus aureus (MRSA) respiratory infection in patients with cystic fibrosis has increased dramatically over the last decade. Epidemiologic evidence suggests that persistent infection with MRSA may result in an increased rate of decline in FEV1 and shortened survival. Treatment of MRSA is a top priority. Inhaled antibiotics offer the advantage of high concentrations of antibiotic at the site of infection (the airway) while minimizing systemic side effects. Vancomycin is a glycopeptide antibiotic that has activity against MRSA. Anecdotal and retrospective peer-reviewed studies have demonstrated that inhaled vancomycin is safe and potentially effective in patients with cystic fibrosis and MRSA airway infection. Data evaluating the pharmacokinetics of vancomycin in sputum are needed before pursuing treatment trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age.
* Confirmed diagnosis of CF based on the following criteria:

  * positive sweat chloride > 60 mEq/liter (by pilocarpine iontophoresis) and/or
  * a genotype with two identifiable mutations consistent with CF or abnormal NPD, and
  * one or more clinical features consistent with the CF phenotype.
* Chronic sputum producer able to spontaneously produce sputum
* FEV1 > 40% of predicted normal for age, gender, and height
* Previous use of any inhaled antibiotics within the last year
* Ability to provide written informed consent
* Ability to adhere to the protocol

Exclusion Criteria:

* Use of inhaled or intravenous vancomycin within two weeks of the study visit
* Known history of intolerance to inhaled vancomycin or inhaled albuterol.
* Known history of hypersensitivity to vancomycin or other glycopeptide antibiotics
* History of sputum culture with Burkholderia cepacia complex in the last two years.
* Pregnancy
* Woman who are lactating and not willing to stop nursing on the day of the study visit and the subsequent 48 hours.
* Current use of oral corticosteroids in doses exceeding the equivalent of 10mg of prednisone a day or 20mg of prednisone every other day.
* Patients not willing to hold other inhaled antibiotics (for example TOBI, Cayston, or Colistin) for at least 2 days prior to the study visit.
* Patients not willing to hold loop diuretics (i.e. furosemide, torsemide, ethacrynic acid) on the morning of the study visit.
* History of ABPA or reactive airways disease that has required treatment within the last year.
* Creatinine greater than 2.0 mg/dL within the last year.
* Oxygen saturation ≤ 92% on room air.
* History of patient reported hearing loss
* Any serious or active medical or psychiatric illness, which in the opinion of the investigator, would interfere with patient treatment, assessment, or adherence to the protocol.
* History of or listed for solid organ or hematological transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01 (Estimated); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | Predose, 5 minutes, one hour, 2 hours, and 6 hours after completion of 250mg of inhaled vancomycin
  Pharmacokinetic analysis will be performed with non-compartmental methods. The area under the curve for sputum vancomycin will be determined.

SECONDARY OUTCOMES:
Change in FEV1% Predicted | 30 minutes
  Change in FEV1% predicted from baseline to 30 minutes after completion of inhaled vancomycin
Change in Patient Symptoms | 6 hours
  Patient's respiratory symptoms and potential side effects from inhaling vancomycin will be queried using a questionnaire prior to inhaling vancomycin, at 15 ±10 minutes, and 4 ± 1 hour after completing inhaled vancomycin.
Change in Sputum Cell Counts | 6 hours
  Change in sputum cell counts (i.e. eosinophils) between baseline and six hours after completion of inhaled vancomycin.
Serum Vancomycin Peak Concentration | 60 minutes
  Serum vancomycin peak concentration 60 minutes after completion of inhaled vancomycin.
Oxygen Saturation | 5 minutes
  Continuous oxygen saturation monitoring to be continued throughout vancomycin inhalation and for 5 minutes after inhalation
Adverse Events | 6 hours
  Information regarding occurrence of adverse events will be captured throughout the study. Duration (start and stop times), severity/grade, outcome, treatment and relation to study medication will be recorded
Maximum Concentration | Predose, 5 minutes, one hour, 2 hours, and 6 hours after completion of 250mg of inhaled vancomycin
  Pharmacokinetic analysis will be performed with non-compartmental methods. The maximum concentration of sputum vancomycin will be determined.
Time to Peak Concentration | Predose, 5 minutes, one hour, 2 hours, and 6 hours after completion of 250mg of inhaled vancomycin
  Pharmacokinetic analysis will be performed with non-compartmental methods. The time to peak concentration for sputum vancomycin will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Elliott C Dasenbrook, MD MHS, Principal Investigator — Case Western Reserve University School of Medicine
Locations (1):
- Rainbow Babies and Children's Hospital, Univeristy Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Dasenbrook EC, Checkley W, Merlo CA, Konstan MW, Lechtzin N, Boyle MP. Association between respiratory tract methicillin-resistant Staphylococcus aureus and survival in cystic fibrosis. JAMA. 2010 Jun 16;303(23):2386-92. doi: 10.1001/jama.2010.791. PMID 20551409
- [Background] Dasenbrook EC, Merlo CA, Diener-West M, Lechtzin N, Boyle MP. Persistent methicillin-resistant Staphylococcus aureus and rate of FEV1 decline in cystic fibrosis. Am J Respir Crit Care Med. 2008 Oct 15;178(8):814-21. doi: 10.1164/rccm.200802-327OC. Epub 2008 Jul 31. PMID 18669817
- [Background] Dasenbrook EC. Update on methicillin-resistant Staphylococcus aureus in cystic fibrosis. Curr Opin Pulm Med. 2011 Nov;17(6):437-41. doi: 10.1097/MCP.0b013e32834b95ed. PMID 21918450
- [Background] Doe SJ, McSorley A, Isalska B, Kearns AM, Bright-Thomas R, Brennan AL, Webb AK, Jones AM. Patient segregation and aggressive antibiotic eradication therapy can control methicillin-resistant Staphylococcus aureus at large cystic fibrosis centres. J Cyst Fibros. 2010 Mar;9(2):104-9. doi: 10.1016/j.jcf.2009.11.009. Epub 2010 Jan 3. PMID 20051329